CLINICAL TRIAL: NCT00347321
Title: Evaluation of Early Percutaneous Tracheostomy in Patients Undergoing Cardiovascular Surgery and Requiring Prolonged Mechanical Ventilation
Brief Title: Early Percutaneous Tracheostomy for Cardiac Surgery (ETOC)
Acronym: ETOC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Christophe AUCAN, Department Clinical Research of Developpement
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P051013
Record Dates: First submitted 2006-06-29; First posted 2006-07-04 (Estimated); Last update posted 2009-12-03 (Estimated); Status verified 2007-03

CONDITIONS: Respiratory Failure; Cardiovascular Surgery
Keywords: Percutaneous tracheostomy; Endotracheal intubation; Mechanical ventilation; Cardiac surgery; Ventilator-free days
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dilatational Percutaneous tracheostomy (Experimental): Dilatational Percutaneous tracheostomy
  Interventions: Procedure: Dilatational Percutaneous tracheostomy

INTERVENTIONS:
Procedure: Dilatational Percutaneous tracheostomy — Dilatational Percutaneous tracheostomy

SUMMARY:
This is a phase III clinical trial comparing early tracheostomy (day 4) versus prolonged endotracheal intubation in ICU patients needing prolonged ventilatory support after cardiovascular surgery.

DETAILED DESCRIPTION:
Background: Prolonged mechanical ventilation (MV> 7 days) is required in less than 10% of patients after cardiovascular surgery but it is associated with high morbidity and mortality.

Several studies conducted in critically ill patients suggested that early percutaneous tracheotomy compared with delayed tracheotomy decreases the length of ventilator dependence and improves outcome. To date, no randomized trial has tested these possible benefits in critically ill patients after cardiac surgery.

Study objectives: A randomized trial has been designed to determine whether early tracheostomy (day 4 after cardiac surgery) in patients still on MV would reduce the number of days under MV, measured by the evaluation of ventilator-free days (VFDs). Secondary objectives are the reduction of mortality, reduction of ICU and hospital length of stay. Evaluation of organ failure evolution, infectious complications, sedation needs, patient comfort and outcome at 3 months will be also considered.

Study hypothesis: The trial will be consider positive if early tracheotomy increases the number VFDs of at least 7 days (mean) evaluated on day 60 after randomisation.

Methods :

Trial : randomized, open, controlled, monocentric Inclusion criteria: see columns below Exclusion criteria: see columns below Randomization: will use a computerised system on day 4 after cardiac surgery Procedures: see columns below Recorded data: demographic characteristics, pre, per and postoperative parameters.

From randomization until ICU discharge (or day 60), a daily chart will be completed.

Judgment criteria: see columns below Sample size and statistical analysis: using Wilcoxon bilateral test with an alpha risk of 5% and a power of 80%, we calculated that 108 patients in each arm would be needed.

Statistical analyses will use standard tests to compare population of the two arms.

ELIGIBILITY:
Inclusion Criteria:

* Are 18 years of age or older
* Have undergone cardiovascular surgery
* Are still on invasive mechanical ventilation on day 4 after surgery
* Have failed the screening test or the spontaneous breathing trial
* Have signed the informed consent (patient or legal representative)

Exclusion Criteria:

* Age less than18
* Pregnant woman
* Intubation more than 48 hours before cardiovascular surgery
* More than 5 days on mechanical ventilation after cardiac surgery
* Artificial heart implantation
* Concomitant neck surgery (carotid)
* Previously tracheostomized
* Major hemorrhagic risk
* Persistence of platelet count less than 50.000/mm3 after platelet transfusion
* Prothrombin time less than 30% despite coagulation factors administration
* Clinical evidence of ongoing infection at the proposed tracheotomy site
* Anatomical deformity of the neck making risky a tracheostomy
* Probability of dying the day of randomization defined by SAPSII more than 80
* Irreversible neurological lesions
* Decision of care limitation
* Prior inclusion in a trial with morbidity-mortality as main judgement criteria
* Previous enrollment in this trial
* Consent refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2006-07; Primary Completion 2009-03 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Number of ventilator-free days defined as the number of days between successful weaning from MV and day 60 after study enrolment. | between successful weaning from MV and day 60 after study enrolment.
VFDs = 0 if the patient dies before 60days. | before 60 days
VFDs= (60- X) : if the patient is successfully weaned from MV within 60 days, where X is the number of days spent receiving MV | during 60 days
VFDs = 0: if the patient requires MV for 60 days or more | during 60 days and after
The trial will be considered positive if early tracheostomy increases the number VFDs of at least 7 days (mean) | at 7 days

SECONDARY OUTCOMES:
Other outcomes will be compared between the two arms: | during the trial
Mortality rate (day 60, in-ICU, in-hospital) | during the 60 days
ICU length of stay | during the trial
Hospital length of stay | during the trial
Duration of MV in survivors | during the trial
Organ failure evolution | during the trial
Infectious complications | during the trial
Early laryngeal and tracheal complications | during the trial
Sedation needs | during the trial
Patient comfort | during the trial
Outcome on day 90 | to 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Jean Louis TROUILLET, MD,, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Institut de Cardiologie - Chu Pitie Salpetriere Ap-Hp, Paris, France

REFERENCES:
- [Derived] Trouillet JL, Luyt CE, Guiguet M, Ouattara A, Vaissier E, Makri R, Nieszkowska A, Leprince P, Pavie A, Chastre J, Combes A. Early percutaneous tracheotomy versus prolonged intubation of mechanically ventilated patients after cardiac surgery: a randomized trial. Ann Intern Med. 2011 Mar 15;154(6):373-83. doi: 10.7326/0003-4819-154-6-201103150-00002. PMID 21403073